CLINICAL TRIAL: NCT04309032
Title: A Randomized Controlled Trial on the Effect of Retrograde Partial Bladder Fill on Time to Discharge and Overall Medical Staff Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hakmin Lee, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1806-474-004
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Retrograde Bladder Fill

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder fill (Experimental): Retrograde bladder filling of 250cc of 0.9% normal saline for irrigation prior to removal of foley catheter
  Interventions: Procedure: retrograde bladder filling with 0.9% normal saline 250cc prior to removal of foley catheter
- No bladder Fill (No Intervention): no filling prior to removal of foley catheter

INTERVENTIONS:
Procedure: retrograde bladder filling with 0.9% normal saline 250cc prior to removal of foley catheter — 0.9% NS 250cc was introduced before foley catheter removed for discharge
  Arms: Bladder fill

SUMMARY:
This study is a randomized controlled trial on the effect of retrograde partial bladder fill on time to discharge in patients who have had urological surgery for BPH, and whether it affects overall medical staff satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Any male patient between ages 20-80 with foley catheter indwelled after urological surgery performed at our institution

Exclusion Criteria:

* Any patient that does not remove foley catheter at discharge

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Time to void | 1day
  time from foley catheter removal to actual initial voiding
Time to discharge | 1day
  time from foley catheter removal to actual discharge
Medical staff satisfaction | 1year
  Medical staff satisfaction discomfort/satisfaction with overall process based on a Likert scale (5)
Patient satisfaction | 1day
  patient discomfort/satisfaction with overall process based on a Likert scale (5)

CONTACTS AND LOCATIONS:
Overall Officials: Hakmin Lee, M.D., Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No